CLINICAL TRIAL: NCT04688905
Title: Diagnosestellung Der Herzinsuffizienz Mit Erhaltener Ejektionsfraktion Bei Patienten Mit Unklarer Belastungsdyspnoe - Validierung Gegen Den Invasiven Goldstandard (Diagnose-HFpEF)
Brief Title: Diagnosing Heart Failure With Preserved Ejection Fraction in Patients With Unexplained Dyspnea (Diagnose-HFpEF)
Status: Active, not recruiting | Type: Observational
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Rolf Wachter, Professor, University of Leipzig
Other Study IDs: 283/20
Record Dates: First submitted 2020-12-04; First posted 2020-12-30 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Dyspnea
MeSH Terms: conditions — Dyspnea | interventions — Coronary Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Approximately 40 ml of blood will be drawn for the conduction of hemogram, sodium, potassium, creatine, eGFR, urea, coagulation, TSH, CK, high-sensitivity troponin T, NT-proBNP, HbA1c, lipids, iron status as well as biobanking (at -80°C) for 15 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dyspnea explained by heart failure with preserved ejection fraction: All patients fulfilling invasive criteria for heart failure with preserved ejection fraction
  Interventions: Diagnostic Test: Invasive hemodynamics of left ventricle via conductance catheter at rest, with exercise and with temporary vena cava occlusion
- Dyspnea not explained by heart failure with preserved ejection fraction: All patients not fulfilling invasive criteria for heart failure with preserved ejection fraction
  Interventions: Diagnostic Test: Invasive hemodynamics of left ventricle via conductance catheter at rest, with exercise and with temporary vena cava occlusion

INTERVENTIONS:
Diagnostic Test: Invasive hemodynamics of left ventricle via conductance catheter at rest, with exercise and with temporary vena cava occlusion — Invasive hemodynamics of left ventricle will be done by the conductance method. Left ventricular stiffness constant will be obtained by temporary vena cava occlusion. Right heart catherization will be done by pulmonary artery catherization and cardiac output will be estimated by thermodilution and Fick´s method.
  Other Names: Cardiac MRI at rest; Echocardiography at rest and with exercise; Spiroergometry; 6 minute walking distance; Right heart catherization at rest and with exercise; Coronary angiography (if not performed within the last year)

SUMMARY:
Invasive diagnosis of heart failure with preserved ejection fraction (HFpEF) in patients with unexplained dyspnea NYHA II-III compared to other diagnostic tools

DETAILED DESCRIPTION:
Multiple diagnostic tests, including stress tests and the invasive conduction of left ventricular pressure-volume loops via conductance catheter (as gold standard) will be performed in patients with unexplained dyspnea NYHA II-III in order to identify patients with a heart failure with preserved ejection fraction (HFpEF). The results will be compared to previously reported diagnostic scores such as the H2FPEF and the HFA-PEFF score.

ELIGIBILITY:
Inclusion Criteria:

* dyspnea NYHA II-III
* age 18-90 years
* left ventricular ejection fraction ≥ 50%
* ability to give informed consent

Exclusion Criteria:

* unstable cardiac disease with acute decompensation
* documented former LVEF ≤ 40%
* heart valve disease with medium or high grade insufficiency or stenosis
* coronary heart disease with hemodynamically relevant coronary stenosis
* specific cardiomyopathia
* acute or chronic cardiac inflammation (myocarditis, pericarditis)
* former heart transplantation
* relevant pulmonary disease (e.g. COPD) assumably causing the dyspnea
* FEV1/VC < 70%
* hemoglobin < 5 mmol/l
* pregnant or nursing women
* contraindication for one of the diagnostic tests

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unexplained dyspnea NYHA II-III
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
HFpEF-positive patients | Within one day
  Percentage of patients with invasively diagnosed heart failure with preserved ejection fraction

SECONDARY OUTCOMES:
H2FPEF score | Within two days
  Difference in H2FPEF score in patients with approved and excluded HFpEF (BMI > 30 kg/m²: 2 points, 2 or more antihypertensive medicines: 1 point, atrial fibrillation: 3 points, pulmonary hypertension: 1 point, age > 60 years: 1 point, E/E' > 9: 1 point. Sum: 0-9 points with rising probability of HFpEF with increasing score)
HFA-PEFF score | Within two days
  Difference in HFA-PEFF score in patients with approved and excluded HFpEF (0-2 points regarding functional, morpholigical and biomarker parameters. Sum: 0-6 points; 0-1 points:exclusion of HFpEF, 2-5 points: further diagnostic (stress test or invasive) required, 5-6 points: HFpEF diagnosed.
Difference in DPVQ (echocardiographic) | Within two days
  Diastolic pressure-volume quotient (DPVQ) (at rest and under exertion) in patients with approved and excluded HFpEF
Difference in E/E' (echocardiographic) | Within two days
  E/E' (at rest and under exertion) in patients with approved and excluded HFpEF
Difference in GLS (echocardiographic) | Within two days
  Global longitudinal strain (at rest and under exertion) in patients with approved and excluded HFpEF
Difference in MRI parameters | Within two days
  Fibrosis (using late gadolinium enhancement and T1-Mapping) in patients with approved and excluded HFpEF
Difference in pulmonary artery pressure (right heart catheter) | Within two days
  Pulmonary artery pressure at rest and under exertion in patients with approved and excluded HFpEF
Difference in wedge pressure (right heart catheter) | Within two days
  Wedge pressure at rest and under exertion in patients with approved and excluded HFpEF
Difference in DPVQ (echocardiographic) after one year | 1 year
  Diastolic pressure-volume quotient (DPVQ) at rest in patients with approved and excluded HFpEF after one year
Difference in E/E' (echocardiographic) after one year | 1 year
  E/E' at rest in patients with approved and excluded HFpEF after one year
Difference in GLS (echocardiographic) after one year | 1 year
  Global longitudinal strain at rest in patients with approved and excluded HFpEF after one year

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Available upon reasonable scientific request.

REFERENCES:
- [Result] Gessner R, Hubner AC, Stobe S, Rudolph UM, Unger L, Schmeisser A, Steendijk P, Uhe T, Stegmann T, Lavall D, Hagendorff A, Laufs U, Wachter R. Diagnosing HFpEF in Patients With Unexplained Dyspnea by Using Invasive Left Ventricular Pressure-Volume Loops. J Card Fail. 2025 Nov;31(11):1661-1671. doi: 10.1016/j.cardfail.2025.09.010. PMID 41233022